CLINICAL TRIAL: NCT02466919
Title: Strategy on the Increment of H. Pylori Eradication Rate and Investigating the Gastric Pathology and Antimicrobial Resistance in Diabetic Patients
Brief Title: Study of Levofloxacin-based Concomitant Therapy for H. Pylori Eradication in Diabetic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chung-Tai Wu (Other)
Collaborators: Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Sponsor-Investigator, Chung-Tai Wu, National Cheng-Kung University Hospital, National Cheng-Kung University Hospital
Organization: National Cheng-Kung University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOHW103-TDU-B-211-113002
Record Dates: First submitted 2015-05-17; First posted 2015-06-09 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori
MeSH Terms: interventions — Pantoprazole; Amoxicillin; Metronidazole; Levofloxacin; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levofloxacin-based concomitant (Experimental): Pantoprazole 40 mg BID day1~day10 Amoxicillin 1000 mg BID day1~day10 Metronidazole 500 mg BID day1~day10 Levofloxacin 500 mg QD day1~day10
  Interventions: Drug: Pantoprazole; Drug: Amoxicillin; Drug: Metronidazole; Drug: Levofloxacin
- Sequential (Active Comparator): Pantoprazole 40 mg BID day1~day10 Amoxicillin 1000 mg BID day1~day5 Metronidazole 500 mg BID day6~day10 Clarithromycin 500 mg BID day6~day10
  Interventions: Drug: Pantoprazole; Drug: Amoxicillin; Drug: Metronidazole; Drug: Clarithromycin

INTERVENTIONS:
Drug: Pantoprazole — H. pylori eradication therapy
  Other Names: Pantoloc
Drug: Amoxicillin — H. pylori eradication therapy
Drug: Metronidazole — H. pylori eradication therapy
  Other Names: Flagyl
Drug: Levofloxacin — H. pylori eradication therapy
  Other Names: Cravit
  Arms: Levofloxacin-based concomitant
Drug: Clarithromycin — H. pylori eradication therapy
  Other Names: Klaricid
  Arms: Sequential

SUMMARY:
The study aims to evaluate H. pylori eradication rate in diabetic patients by using novel 10-day levofloxacin-based concomitant therapy compared with conventional 10-day sequential therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with Helicobacter pylori infection

Exclusion Criteria:

* Pregnancy or physically poor performance status
* Patients with contraindication for upper endoscopy
* Severe coagulopathy for endoscopic biopsy
* Chronic kidney disease (eGFR < 50) or end stage renal disease
* Known allergy to interventional drugs
* Previous eradication failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2014-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | 1-4 months after eradication therapy
  C13-UBT to confirm the H. pylori eradication

SECONDARY OUTCOMES:
Acute inflammatory score | 1-4 weeks after gastric tissue obtained by upper endoscopy
  Gastric tissue obtained from antrum (2 pieces), body (2 pieces) and cardia (1 piece) were scoring by modified Sydney system and specific staining. Acute inflammatory score (AIS) can be assessed by the sum of these five pathologic tissues
Chronic inflammatory score | 1-4 weeks after gastric tissue obtained by upper endoscopy
  Chronic inflammatory score (CIS) can be assessed by the sum of these five pathologic tissues
H. pylori density score | 1-4 weeks after gastric tissue obtained by upper endoscopy
  H. pylori density score (HPDS) can be assessed by the sum of these five pathologic tissues
Intestinal metaplasia | 1-4 weeks after gastric tissue obtained by upper endoscopy
  Presence of intestinal metaplasia can be evaluated from these five pathologic tissues
Spasmolytic polypeptide expressing metaplasia | 1-4 weeks after gastric tissue obtained by upper endoscopy
  Presence of spasmolytic polypeptide expressing metaplasia can be evaluated from these five pathologic tissues by special TFF-2 stains
H. pylori resistance panel | 1-4 weeks after H. pylori culture obtained by upper endoscopy
  E-test evaluation for antibiotic (amoxicillin, metronidazole, clarithromycin, tetracycline and levofloxacin) resistance

CONTACTS AND LOCATIONS:
Overall Officials: Yao-Jong Yang, PhD, Principal Investigator — National Cheng-Kung University Hospital

REFERENCES:
- [Derived] Yang YJ, Wu CT, Ou HY, Lin CH, Cheng HC, Chang WL, Chen WY, Yang HB, Lu CC, Sheu BS. Male non-insulin users with type 2 diabetes mellitus are predisposed to gastric corpus-predominant inflammation after H. pylori infection. J Biomed Sci. 2017 Oct 30;24(1):82. doi: 10.1186/s12929-017-0389-x. PMID 29082856
- [Derived] Yang YJ, Wu CT, Ou HY, Lin CH, Cheng HC, Chang WL, Chen WY, Yang HB, Lu CC, Sheu BS. Ten days of levofloxacin-containing concomitant therapy can achieve effective Helicobacter pylori eradication in patients with type 2 diabetes. Ann Med. 2017 Sep;49(6):479-486. doi: 10.1080/07853890.2017.1294761. Epub 2017 Mar 7. PMID 28266875